CLINICAL TRIAL: NCT07273565
Title: Feasibility of Comparing Microwave Images and Mammograms in Patients Recalled for Follow-up Breast Imaging
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Pureform Radiology (Unknown); Wave View Imaging Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HREBA.CC-25-0255
Record Dates: First submitted 2025-11-18; First posted 2025-12-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Breast - Female
Keywords: women; mammography; recall; breast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WVI-MIS-02-2025 (Experimental): A single arm study in which the collected microwave data is compared against available clinical data.
  Interventions: Device: WVI-MIS-02-2025

INTERVENTIONS:
Device: WVI-MIS-02-2025 — Microwave scans

SUMMARY:
The goal of this clinical trial is to measure the electrical properties of breast tissues using microwave technology and to compare these collected measurements to clinical information in mammograms for women that have been recalled for follow-up breast imaging. The main questions it aims to answer are:

1. Can the breast area and plate separation in the microwave scan be compared to mammogram data to assess similarity in breast positioning and the feasibility of image registration?
2. Can the distribution of electrical properties specifically glandular tissue distribution in the microwave image be compared to that observed in the mammogram?
3. Can the characteristics of the microwave image in the localized region corresponding to an identified anomaly in the mammogram be examined?

Study participants will be scanned with the Wave View microwave scanner on the same day as their follow-up breast imaging appointment. Each breast will be scanned up to 3 times with the scanner oriented in both the horizontal position and oriented at 45 degrees. Study participants will also be asked to fill out three surveys, one relating to breast health and the other two relating to their scanning experience.

DETAILED DESCRIPTION:
A new approach to imaging that uses low-power microwaves to scan the breast has been developed. Since the imaging system uses low power, there is no risk of tissue heating. The imaging system places the sensors in contact with the breast tissue. The research team at the University of Calgary has previously developed microwave imaging systems that have been tested on healthy volunteers and breast cancer patients. A group of healthy volunteers were repeatedly scanned to evaluate the consistency of the imaging approach. Another study involved scanning breast cancer patients before each round of neoadjuvant chemotherapy. The information collected from experiences scanning volunteers and patients have been reviewed and translated into a next-generation imaging system design. Aspects of this system have been further improved by Wave View Imaging, which is a company formed by members of the University's research team.

The proposed study involves collecting electrical property measurements of breast tissues and comparing these measurements to clinical information in mammograms. The investigators also aim to compare regions of interest in the microwave scans with regions of interest in the mammograms. This includes regions dominated by fibroglandular tissues, as well as regions of interest that correspond to anomalies identified in the mammograms.

The plan is to scan both breasts of up to 20 volunteers that have been recalled for follow-up breast imaging. Each volunteer will participate in a single scanning session during their follow-up appointment. Breast tissue composition will be compared with the microwave properties and registration of mammograms with microwave images will be performed for a more detailed comparison.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* 18-74 years of age
* Able to provide informed consent
* Had a screening mammogram within the previous 6 weeks
* Recalled for additional breast imaging due to BIRADS 3 or 4 findings.

Exclusion Criteria:

* Participants who have not received a mammogram
* Participants who are currently undergoing breast cancer treatment or have had treatment in the past 6 months
* Participants with breast implants
* Participants who are pregnant or breastfeeding
* Participants with active breast skin infections
* Participants with nipple piercings (unless they are removed prior to scanning)
* Participants with an implanted electronic device
* Participants with physical limitations that prevent them from placing their breasts inside the Wave View scanner.

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of electrical properties of breast tissues in microwave images | 12 months
  The average electrical properties of the Wave View image will be calculated (relative permittivity and attenuation). The average properties of the right and left breasts will be compared. The average properties of the craniocaudal (CC) and mediolateral oblique (MLO) views will also be compared for both breasts.

SECONDARY OUTCOMES:
Examine the similarity in plate separation between mammography and Wave View scans | 12 months
  The separation between the plates contacting the breast will be compared between the two modalities. This comparison provides an initial indication of the volume of breast tissue in the scanner.
Breast area | 12 months
  The breast area on the mammogram will be compared to the breast area on the Wave View scan. The breast area in the Wave View image will be calculated, while the breast area on the mammogram is available from automated image analysis reports.
Examine the similarity between glandular tissue distribution on mammograms and electrical property images obtained with the Wave View scanner. | 12 months
  The microwave image will be overlayed on the mammogram to provide initial insight on glandular tissue distribution via visual inspection. The images will be registered based on the outline of the breast. If the breast areas are found to differ, deformable registration techniques will be applied. Higher intensity regions representing glandular tissues will be identified in both images via image filtering and segmentation. These regions will be compared with metrics such as the Dice coefficient. In addition, the area of the higher intensity region will be compared with the overall area of the breast image, similar to the method used to calculate the percentages used in breast density analysis.
Examine how closely the presence of responses in Wave View scans correspond to anomalies detected on mammograms | 12 months
  Localized regions in the Wave View image that correspond to locations of anomalies on the mammogram will be identified based on the registered images. The average properties of these regions will be compared with the average properties of a region in the same breast, as well as in the contralateral breast.
Estimate of breast composition | 12 months
  Pureform Radiology uses a breast density tool to automatically calculate the volume of the breast and glandular tissue, as well as the percentage density and density category (A, B, C, D). Microwave properties are expected to be greater with greater breast densities.To compare electrical properties to breast density, average electrical properties of each microwave scan will be plotted against the corresponding percent density.

CONTACTS AND LOCATIONS:
Locations (1):
- Pureform Radiology, Calgary, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] C. M. Butterworth, P. Mojabi, and E. C. Fear, "Quantifying Consistency of Microwave Breast Imaging: Laser Scanning for Assessing Breast Volume and Shape," IEEE Journal of Electromagnetics, RF and Microwaves in Medicine and Biology, pp. 1-9, 2025, doi: 10.1109/JERM.2025.3531693
- [Result] Mojabi P, Bourqui J, Lasemiimeni Z, Grewal B, Fear E. Microwave Imaging for Breast Cancer Detection: Performance Assessment of a Next-Generation Transmission System. IEEE Trans Biomed Eng. 2025 Jun;72(6):1787-1799. doi: 10.1109/TBME.2024.3521410. PMID 40031671
- [Result] Wang Z, Mojabi P, Price S, Lasemiimeni Z, Besler B, Bourqui J, Deutscher D, Besler B, Shen H, Docktor B, Tsang RY, Fear E. Reproducibility of Microwave Breast Imaging: Analysis of Regular Scans of a Group of Volunteers. IEEE Trans Biomed Eng. 2025 May;72(5):1562-1571. doi: 10.1109/TBME.2024.3512572. Epub 2025 Apr 22. PMID 40030750
- [Result] Mojabi P, Bourqui J, Fear E. Fast 3D Breast Imaging With a Transmission-Based Microwave System. IEEE Trans Med Imaging. 2025 May;44(5):2206-2217. doi: 10.1109/TMI.2025.3527916. Epub 2025 May 2. PMID 40030952
- [Result] Smith K, Bourqui J, Wang Z, Besler B, Lesiuk M, Roumeliotis M, Quirk S, Grendarova P, Pinilla J, Price S, Docktor B, Fear E. Microwave imaging for monitoring breast cancer treatment: A pilot study. Med Phys. 2023 Nov;50(11):7118-7129. doi: 10.1002/mp.16756. Epub 2023 Oct 6. PMID 37800880
- [Result] Smith, K., et al. "Microwave Imaging of the Breast: Consistency of Measurements Over Time." IEEE Journal of Electromagnetics, RF and Microwaves in Medicine and Biology, vol. 6, no. 1, 2022, pp. 61-67, https://doi.org/10.1109/JERM.2021.3099014. . : . .